CLINICAL TRIAL: NCT02029001
Title: A Two-period, Multicenter, Randomized, Open-label, Phase II Study Evaluating the Clinical Benefit of a Maintenance Treatment Targeting Tumor Molecular Alterations in Patients With Progressive Locally-advanced or Metastatic Solid Tumors
Brief Title: Adapting Treatment to the Tumor Molecular Alterations for Patients With Advanced Solid Tumors: MyOwnSpecificTreatment
Acronym: MOST plus
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Leon Berard (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ET12-081; 2012-004510-34 (EudraCT Number)
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Malignant Solid Neoplasms
Keywords: Solid tumor; Recurrent/metastatic; Personalized medicine; Genomic alteration; Targeted therapy; Nilotinib; Everolimus; Sorafenib; Lapatinib; Pazopanib; Olaparib; Immunotherapy; Durvalumab; Tremelimumab
MeSH Terms: conditions — Neoplasm Metastasis | interventions — nilotinib; BID protein, human; Everolimus; Cohort Studies; Sorafenib; Lapatinib; pazopanib; olaparib; durvalumab; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Maintenance treatment (Experimental): Patients will continue targeted treatment matching the molecular alterations identified in their tumor
  * for a maximum of 136 weeks starting from the date of patient's first study drug intake following inclusion or a discontinuation criteria (unacceptable toxicity, interruption of study drug more than 28 days, documented on-treatment disease progression, patient decision, investigator decision, pregnancy) is met for nilotinib, everolimus, sorafenib, lapatinib, pazopanib, olaparib.
  * until loss of clinical benefit, or until a permanent study drug discontinuation criteria is met (unacceptable toxicity, interruption of study drug more than 28 days, documented on-treatment disease progression, patient decision, investigator decision, pregnancy) or for up to 2 years duration for patients with CR/PR/SD with the possibility of rechallenge in case of PD after IT cessation for durvalumab + tremelimumab
  Interventions: Drug: Nilotinib (400 mg BID); Drug: Everolimus (10 mg QD); Drug: Sorafenib (400 mg BID); Drug: Lapatinib (1500 mg QD); Drug: Pazopanib (800 mg QD); Drug: Olaparib (300 mg BID); Combination Product: Durvalumab + Tremelimumab
- Arm B:Interruption of targeted treatment (No Intervention): Targeted treatment received during induction period will be discontinued until a first documented off-treatment disease progression occurs. At progression, treatment reintroduction may be proposed to the patient (left at the investigator's appreciation, and upon patient approval).
  Treatment may be continued until on-treatment disease progression, unacceptable toxicity or for a maximum of 136 weeks from the date of patient's first study drug intake following inclusion for nilotinib, everolimus, sorafenib, lapatinib, pazopanib, olaparib or until loss of clinical benefit, or until a permanent study drug discontinuation criteria is met for durvalumab + tremelimumab.
  If the investigator considers that the treatment cannot be safely reintroduced (regarding patient's condition and/or laboratory results), the patient will be withdrawn from study.

INTERVENTIONS:
Drug: Nilotinib (400 mg BID) — Patient with advanced pigmented villonodular synovitis and tumors with mutations of ABL1, KIT, PDGFRA, PDGFRB, DDR1, DDR2, CSF1R, or amplification/translocation of the genes and/or of the ligands.
  Other Names: Open cohort
  Arms: Arm A: Maintenance treatment
Drug: Everolimus (10 mg QD) — Patients whose tumor harbors mutations or amplification of the PIK3CA, PIK3R1, AKT1, AKT2, mTOR, RICTOR, RAPTOR genes, or with TSC1, TSC2 or PTEN loss (defined as complete loss of both gene copies OR loss of one copy + mutation on the other copy or loss of one copy + loss of expression using immunohistochemistry).
  Other Names: Closed cohort
  Arms: Arm A: Maintenance treatment
Drug: Sorafenib (400 mg BID) — Patients whose tumor harbors mutations of VEGFR1-3, PDGFRB, FLT3, BRAF (other than V600 mutations), CRAF, HRAS, KRAS or RET or amplification/translocation of the genes and/or of the ligands.
  Other Names: Closed cohort
  Arms: Arm A: Maintenance treatment
Drug: Lapatinib (1500 mg QD) — Patients whose tumor harbors mutations or amplifications of HER2
  Other Names: Closed cohort
  Arms: Arm A: Maintenance treatment
Drug: Pazopanib (800 mg QD) — Patients whose tumor harbors mutations of VEGFR1-3, PDGFRA, PDGFRB or KIT* or amplification /translocation of the genes and/or of the ligands.
  Other Names: Closed cohort
  Arms: Arm A: Maintenance treatment
Drug: Olaparib (300 mg BID) — ATM, BAP1 et BRIP1 Mutation only if double hit documented; BRCA2, BRCA1, RAD51C, PALB2, RAD51D Mutation; BRCA1, BRCA2, ATM and BAP1 Loss; BRCA1, BRCA2, ATM and BAP 1 : mutation and heterozygote deletion. except for patients eligible to olaparib's available labels and reimbursements in France.
  NOTE : only prostate cancer with RECIST 1.1 evaluable disease are eligible until the French price and reimbursement
  Other Names: Open cohort
  Arms: Arm A: Maintenance treatment
Combination Product: Durvalumab + Tremelimumab — Any molecular types of tumor (which are known to be immunogenic or with high mutation load), except lung, urothelial and head and neck or CNS tumors, or patients who fulfill conditions to receive any other MTT of the MOST Plus study.
  Other Names: Open cohort
  Arms: Arm A: Maintenance treatment

SUMMARY:
The MOST Plus study is a two-period phase II clinical trial, conducted in patients with all types of progressive solid tumors after at least 1 prior systemic treatment regimen for advanced disease (in the absence of a validated second line therapy).

The main goal of this study is to evaluate for these patients the clinical benefit of a maintenance treatment in patients with stable disease (SD) after induction treatment with a selected therapy (Molecular Targeted Therapy (MTT) or with SD, partial response (PR) or complete reponse (CR) with Immunotherapy (IT)).

For MTT, the first period of this trial (induction period) will enable to establish whether the identification of genomic alterations in genes encoding for "actionable" targets in the tumor cells, regardless of the histological subtype, can be used to select efficient treatment targeting the pathway activated by the mutation.

For Immunotherapy, induction period with durvalumab + tremelimumab is expected to be an innovative therapy for an efficient tumor control and may allow to identify types of cancer or molecular types of cancer that are more receptive to immunotherapy.

For all treatments, the second period (maintenance period) will use a randomized design to evaluate the clinical benefit of a maintenance treatment with the targeted therapy or immunotherapy selected based on tumor molecular profile in patients treated by MTT with SD and in patients treated by IT with SD, PR or CR.

Each patient enrolled will receive the matching targeted therapy during 12 weeks (MTT) or 52 weeks (IT). At the end of this induction period:

MTT cohorts :

* patients with a tumor response (CR: complete response or PR: partial response) will continue the targeted therapy,
* patients in progression will discontinue the targeted therapy and will be withdrawn from study and oriented towards standard treatments
* patients with a stable disease at 12 weeks will be randomized in order to determine if they continue or stop the therapy.

IT cohort :

- patients with SD, PR or CR at 52 weeks will be randomized in order to determine if they continue or stop the therapy.

For each MTT treatment group: ~80 patients treated in the first step (induction period), 50 patients randomized in the second step (maintenance period, 25 patients per arm).

For IT treatment group: ~125 patients treated in the first step (induction period), 50 patients randomized in the second step (maintenance period, 25 patients per arm).

In total (for 7 treatment groups): ~ 900 patients treated in the induction period and 350 patients randomized in maintenance period.

ELIGIBILITY:
Inclusion Criteria:

I1. Male or female patient ≥ 18 years of age.

I2. Histologically or cytologically confirmed diagnosis of metastatic or locally advanced and unresectable solid tumor of any type, except for Nilotinib cohort: only pigmented villonodular synovitis are eligible, not amenable to curative treatment. Concerning primitive tumors of the central nervous system (CNS), all histological types of malignant tumors (including parenchymal and meningeal tumors) are eligible (except for IT).

I3. Documented disease progression at the time of study entry.

I4. At least one prior systemic treatment regimen for locally advanced or metastatic disease - except for Nilotinib cohort : patients can be treated with Nilotinib in first line systemic treatment.

Patients who are candidates for a validated second line treatment regimen are not eligible for the study. For patients with a primitive CNS tumor, the absence of other therapeutic options must be validated by the reference committee for the patient's pathology before inclusion. As there is no prior systemic treatment regimen available for locally advanced or metastatic PEComa, these tumors are eligible for a MTT treatment in first line of their advanced or metastatic disease. No previous treatment by immune checkpoint inhibitors (anti-PD1/PDL1, anti-CTLA4, anti-LAG3 etc.) is allowed for IT group.

I5. Patient with measurable disease, defined as at least one lesion that can be accurately measured on CT-scan or MRI according to RECIST 1.1.

I6. A multidisciplinary molecular board must have recommended one of the investigational MTT available in the study after review of a tumor (or blood for pazopanib, olaparib and immunotherapy cohorts) molecular profiling previously established from a biopsied lesion and/or primitive tumor, and/or from a liquid biopsy, respectively (for pazopanib, olaparib and immunotherapy cohorts).

I7. The MTT recommended by the multidisciplinary molecular board after the review of tumor or blood molecular profile is not approved and reimbursed in France for the disease affecting the patient in the same label.

I8. Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.

I9. Adequate organ system function as assessed by the following minimal laboratory requirements :

* Absolute neutrophil count (ANC) ≥ 1 x 109/L (for pazopanib and olaparib: ≥ 1.5 x 109/L)
* Platelets ≥ 100 x 109/L
* Hemoglobin ≥ 9 g/dL. Transfusion is not allowed within 7 days of screening assessment. (For olaparib: Hemoglobin ≥ 10 g/dL. Transfusion is not allowed within 28 days of screening assessment, no features suggestive of myelodysplastic syndrome (MDS)/Acute myeloid leukemia (AML) on peripheral blood smear within the 28 days)
* For pazopanib: activated partial thromboplastin time (aPTT) ≤ 1.2x Upper limit of normal (ULN) and prothrombin time (PT) or international normalized ratio (INR) ≤ 1.2x ULN; Subjects receiving anticoagulant therapy are eligible if their INR is stable and within the recommended range for the desired level of anticoagulation.
* Aspartate Aminotransferase (AST) and alanine transaminase (ALT) ≤ 3x ULN in the absence of liver metastases (≤ 5x ULN for patients with liver involvement of their cancer) and total bilirubin ≤ 1.5x ULN. (for pazopanib: AST and ALT ≤ 2.5x ULN; concomitant elevations in bilirubin and AST or ALT above 1x ULN are not permitted; for olaparib and IT: AST and ALT ≤ 2.5x ULN in the absence of liver metastases (≤ 5x ULN for patients with liver involvement of their cancer) and total bilirubin ≤ 1.5x ULN.).
* Serum creatinine ≤ 1.5x ULN or creatinine clearance ≥ 50 mL/min (calculated by Cockcroft-Gault formula, or modification of diet in renal disease (MDRD) formula for patients older than 65 years) (for pazopanib: creatinine clearance ≥ 30 mL/min; for olaparib : creatinine clearance ≥ 51 mL/min; for IT : creatinine clearance ≥ 40 mL/min )
* For pazopanib: Urine Protein to Creatinine ratio (UPC) <1; if UPC ≥1, 24-hour urine protein must be <1g (use of urine dipstick for renal function assessment is not acceptable).
* Corrected QT (QTc) interval ≤ 450 msecs (≤ 480 msecs if recommended MTT has no known effect on QT interval) on screening ECG, within 14 days prior to C1D1 (for olaparib : QTc < 470 msec on 2 or more time points within a 24 hour period on screening ECG, within 7 days prior to C1D1).

I10. Life expectancy of at least 4 months.

I11. Specific toxicities related to any prior anti-cancer therapy must have resolved to grade ≤1 (defined by the NCI-CTCAE v4.03) except for alopecia, vitiligo and fatigue. Grade 2 neutropenia or anemia is accepted.

I12. Women of childbearing potential must have a negative pregnancy test performed within 3 days prior to study treatment start. A positive urine test must be confirmed by a serum pregnancy test.

I13. Women of childbearing potential (entering the study after a confirmed menstrual period and who have a negative pregnancy test) and men of reproductive potential must agree, if sexually active, to use two methods of medically acceptable forms of contraception during the study and for at least 8 weeks following the last treatment intake. (for olaparib : during the study and for at least 6 months for women and 3 months for men following the last treatment intake; for IT : during the study and for at least 3 months following the last treatment intake). Refrain from breastfeeding (for nilotinib cohort : not breast-feed for at least two weeks after the last dose of nilotinib) and egg cell donation. Males should not donate sperm during or for 3 months after treatment I14. Signed and dated informed consent document indicating that the patient has been informed of all the pertinent aspects of the trial prior to enrollment.

I15. The patient must be affiliated to the French social security system.

I16. The recommended study treatment must have been approved by the medical staff of the Steering committee.

I17. Patient should be able and willing to comply with study visits and procedures as per protocol.

I18. Patient must fulfill ALL following conditions (criteria only applicable for Durvalumab + Tremelimumab cohort):

* Availability of a pre-treatment sample of primary tumor (only formalin-fixed paraffin-embedded (FFPE) block with sufficient material) and presence of at least one biopsiable tumor lesion for on-treatment biopsy,
* Weight > 50 Kg,
* Patient with a maximum of 2 prior lines of treatment at time of C1D1 for their metastatic or locally advanced.

Exclusion Criteria:

Patients eligible for this study must not meet any of the following criteria:

E1. Previous treatment in advanced phase with an investigational therapy inhibiting the same target proteins as this recommended for the study.

E2. Any contra-indication to receive the recommended MTT, including known or suspected hypersensitivity to compounds of similar chemical or biologic composition as the active substance, or to any of the excipients.

E3. For nilotinib, sorafenib, pazopanib, lapatinib and olaparib: Patient with hypokalemia (< Lower Limit of Normal) or known history of congenital long QT syndrome (QT interval prolongation).

E4. Prior malignancy or presence of any other active malignancy. Subjects who have had another malignancy and have been disease-free for 5 years, or subjects with a history of completely resected non-melanomatous skin carcinoma or successfully treated in situ carcinoma are eligible.

E5. Patient who have had major surgery or trauma within 28 days prior to first dose of investigational product. Patient must have recovered from any effects of any major surgery.

E6. Patient with symptomatic or uncontrolled CNS metastatic involvement of his/her cancer, unless the patient have stable neurological function without evidence of CNS progression within 12 weeks prior to study entry and does not require treatment with enzyme-inducing anticonvulsants or steroids. Patients with a primitive tumor of the CNS are not eligible to IT and if one of the following conditions is fulfilled:

* Alteration of cognitive functions impeding the patient's comprehension of study and the provision of informed consent by the patient himself/herself.
* Need for supportive care treatment(s) interfering with study treatment.

E7. Treatment with any of the following anti-cancer therapies prior to the first dose of study treatment: radiation therapy (for olaparib : within 3 weeks or 5 half-lives of a drug whichever is longer), surgery or tumor embolization within 14 days prior to the first dose of study treatment OR immunotherapy within 28 days (except for IT : patient already treated with an immunotherapy are excluded) OR chemotherapy (for olaparib : within 3 weeks or 5 half-lives of a drug whichever is longer), biologic therapy, investigational therapy or hormonal therapy within 14 days or 5 half-lives of a drug (whichever is longer). Palliative radiotherapy is authorized only if the irradiated field does not include target lesions. Patient already treated with with immune checkpoint inhibitors (anti-PD1/PDL1, anti-CTLA4, anti-LAG3 etc.) are excluded.

E8. Administration of any non-oncologic investigational agent within 30 days or 5 half-lives (whichever is longer) prior to receiving the first dose of study treatment.

E9. For oral treatment : Patient with any condition that impairs their ability to swallow and retain tablets and may affect the absorption of the investigational product are excluded.

E10. For pazopanib: Clinically significant gastrointestinal abnormalities that may increase the risk for gastrointestinal bleeding including, but not limited to:

* Active peptic ulcer disease
* Known intraluminal metastatic lesion(s) with risk of bleeding
* Inflammatory bowel disease or other gastrointestinal conditions with increased risk of perforation
* History of abdominal fistula, gastrointestinal perforation, or intra abdominal abscess within 28 days prior to beginning study treatment.

E11. For pazopanib and IT: Evidence of active bleeding or bleeding diathesis. E12. For pazopanib: Known endobronchial lesions and/or lesions infiltrating major pulmonary vessels that increase the risk of pulmonary hemorrhage.

* Lesions infiltrating major pulmonary vessels (contiguous tumour and vessels) are excluded; however, the presence of a tumor that is touching, but not infiltrating (abutting) the vessels is acceptable.
* Large protruding endobronchial lesions in the main or lobar bronchi are excluded; however, endobronchial lesions in the segmented bronchi are allowed.
* Lesions extensively infiltrating the main or lobar bronchi are excluded; however, minor infiltrations in the wall of the bronchi are allowed.

E13. For pazopanib: Recent hemoptysis.

E14. Any clinically significant and/or uncontrolled medical disease that could compromise the patient's ability to tolerate study treatment or would likely interfere with study procedures or results. These conditions include but are not limited to:

* Active clinically serious bacterial or fungal infection
* History of uncontrolled or significant cardiac disease within the past 6 months: left ventricular ejection fraction (LVEF) < 50%, congestive cardiac failure, active ischemic heart disease, ventricular arrhythmia, myocardial infarction within 1 year, unstable angina pectoris, cardiac surgery. (except for Nilotinib, all patients with uncontrolled or significant cardiac disease are excluded)
* Patients with cerebrovascular accident (including transient ischemic attack), pulmonary embolism or untreated deep venous thrombosis (DVT) within the past 6 months are not eligible for pazopanib treatment group
* Poorly controlled hypertension [for pazopanib: defined as systolic blood pressure (SBP) ≥140 mmHg or diastolic blood pressure (DBP) ≥ 90 mmHg]
* Severely impaired lung function
* Active gastrointestinal tract ulceration
* Acute or chronic uncontrolled liver disease, or severe renal disease
* Uncontrolled diabetes
* Known history of human immunodeficiency virus (HIV) infection, or active viral infection (hepatitis B virus (HBV), hepatitis C virus (HCV)) at the time of study entry and/or requiring anti-viral therapy, or chronic hepatitis B or C. Detection of hepatitis C RNA must be performed before inclusion of patients with a history of HCV infection: patients with a positive result are excluded.
* History of organ allograft or patient taking immunosuppressive treatment.

E15. Patient unable or unwilling to discontinue use of prohibited medications for at least 14 days or 5 half-lives of a drug (whichever is longer) prior to the first dose of study drug and for the duration of the study.

E16. Pregnant or breastfeeding women. E17. Patients with any medical, psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule or evaluations of the study results.

E18. Patient currently treated with drugs that could interfere with study drugs metabolism E19. Patients filling at least one of these criteria are excluded. (Specific to olaparib)

* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patients considered a poor medical risk due to a serious, uncontrolled seizures, uncontrolled medical disorder, non-malignant systemic disease or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent myocardial infarction, unstable spinal cord compression , superior vena cava syndrome, extensive bilateral lung disease on High-resolution computed tomography (HRCT) scan.
* Previous allogenic bone marrow transplant or double umbilical cord blood transplantation and whole blood transfusions in the last 120 days prior to entry to the study (packed red blood cells and platelet transfusions are acceptable) are not allowed.
* Concomitant use of known strong CYP3A inhibitors or moderate CYP3A inhibitors. The required washout period prior to starting olaparib is 2 weeks.
* Concomitant use of known strong or moderate CYP3A inducers. The required washout period prior to starting olaparib is 5 weeks for enzalutamide or phenobarbital and 3 weeks for other agents.
* Patients eligible for olaparib (Lynparza®) in its approved indication in France E20. For IT: Patients filling at least one of these criteria are excluded.
* Patients with lung or urothelial or head and neck cancers or CNS tumors or patients who fulfill conditions to receive one of the investigational therapy of the study
* Current or prior use of immunosuppressive medication within 14 days before the first dose of Durvalumab or Tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10mg/day of prednisone, or an equivalent corticosteroid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 900 (Estimated)
Dates: Start 2014-03 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Induction Progression-Free Rate after induction treatment | 12 weeks for MTT or 52 weeks for IT after initiation of study treatment
  The proportion of patients without documented disease progression within induction period (the first 12 weeks of study treatment or 52 weeks for IT).
Progression-Free Survival (PFS) in both study arms after randomization | 16 weeks after randomisation date
  Measured from the date of randomization until the date of event defined as the first documented progression or death from any cause. Patients with no event at the time of the analysis will be censored at the date of the last available tumor assessment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Over the induction period
  Proportion of patients with complete response (CR) or partial response (PR) as best overall response over the induction period.
Overall survival (OS) | from the date of randomization to the date of death from any cause
Patient's quality of life score (QLQ-C30) in both arms after randomization | At randomization (week 12 for MTT or week 52 for IT), 16 weeks after randomisation (week 28 for MTT or week 68 for IT) and end of study for patient (week 136 for MTT or until up to 130 months after treatment start for IT)
Safety assessment | Over the whole study
  Type, frequency, seriousness and causality of adverse events reported from treatment initiation based on the common toxicity criteria grade (NCI CTC-AE-V4.03)

OTHER OUTCOMES:
Duration of response (exploratory outcome) | Over the whole study
  Measured from the time of first documented response (CR or PR) until the first documented disease progression or death due to underlying cancer, and censored at the date of the last available tumor assessment
Medico-economic evaluation: cost analysis and cost-effectiveness analysis | From randomization until patient's end of study
  Incremental cost-effectiveness ratios (ICERs) will be expressed as:
  * the cost per life year gained;
  * the cost per progression-free year gained.
Progression Free Survival (exploratory outcome) | Through study completion, an average of 1 year
  Measured from the date of the first administration of the treatment until the date of event defined as the first documented progression or death from any cause. Patients with no event at the time of the analysis will be censored at the date of the last available tumor assessment.
Molecular evolution of tumor at progression (for olaparib and durvalumab + tremelimumab groups) | Through study completion, an average of 1 year
  ctDNA analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves BLAY, MD, Principal Investigator — Centre Leon Berard
Locations (7):
- France (7):
  - Institut Bergonié, Bordeaux
  - Centre Leon Berard, Lyon
  - Centre Hospitalier Lyon Sud, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut Curie, Paris
  - Institut de Cancerologie de Strasbourg Europe, Strasbourg
  - Institut Claudius Regaud, Toulouse

REFERENCES:
- [Derived] Tredan O, Toulmonde M, Le Tourneau C, Montane L, Italiano A, Ray-Coquard I, De La Fouchardiere C, Bertucci F, Goncalves A, Gomez-Roca C, You B, Attignon V, Boyault S, Cassier PA, Dufresne A, Tabone-Eglinger S, Viari A, Sohier E, Kamal M, Garin G, Blay JY, Perol D. Sorafenib in Molecularly Selected Cancer Patients: Final Analysis of the MOST-Plus Sorafenib Cohort. Cancers (Basel). 2023 Jun 30;15(13):3441. doi: 10.3390/cancers15133441. PMID 37444551
- See also: MOST study is part of the LyRICAN project, click here to access LyRICAN website — https://www.cancer-lyrican.fr/